CLINICAL TRIAL: NCT01836588
Title: New Gentle Biopsy Method of Cervix Lesions Using Superficial Curettage/Protocol ID: CX-CUR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Deutsche Klinik fuer Diagnostik (Other)
Responsible Party: Principal Investigator, Tim Schellenberg, physician, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CX-CUR
Record Dates: First submitted 2013-03-13; First posted 2013-04-22 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-04

CONDITIONS: CIN; Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

ARMS (2):
- gentle tissue extraction (curettage) (Active Comparator): Object of this study is the evaluation of two different methods of gaining cervical tissue in order to determine whether, and if so in what extent, a CIN is existent. The first method is a cervical biopsy, the second method is a gentle tissue saving curettage of the cervix uteri. Also is to be investigated that the latter method shows a reduction of pain and morbidity after the procedure.
  For this reason the pathological outcome of the two methods will be compared to the result of a conisation, which will be received by the patient to cure their cervical lesions.
  Interventions: Procedure: conventional cervix biopsy
- conventional cervix biopsy (Active Comparator): Object of this study is the evaluation of two different methods of gaining cervical tissue in order to determine whether, and if so in what extent, a CIN is existent. The first method is a cervical biopsy, the second method is a gentle tissue saving curettage of the cervix uteri. Also is to be investigated that the latter method shows a reduction of pain and morbidity after the procedure.
  For this reason the pathological outcome of the two methods will be compared to the result of a conisation, which will be received by the patient to cure their cervical lesions.
  Interventions: Procedure: conventional cervix biopsy

INTERVENTIONS:
Procedure: conventional cervix biopsy — Object of this study is the evaluation of two different methods of gaining cervical tissue in order to determine whether, and if so in what extent, a CIN is existent. The first method is a cervical biopsy, the second method is a gentle tissue saving curettage of the cervix uteri. Also is to be investigated that the latter method shows a reduction of pain and morbidity after the procedure.
  For this reason the pathological outcome of the two methods will be compared to the result of a conisation, which will be received by the patient to cure their cervical lesions.

SUMMARY:
It is to investigate to what extent a gentle tissue extraction of CIN lesions of the cervix will bring the same conclusion than the conventional cervix biopsy, but with less pain and morbidity, after patients were undergoing a conisation in order to treat CIN.

ELIGIBILITY:
Inclusion Criteria:

* Women between 18 and 80
* Karnofsky-Index of 80 and higher
* Cytological suspicious CIN and a colposcopical impression of a major lesion (therapeutical endpoint: conisation)

Exclusion Criteria:

* Former malign disease oft he pelvic organs
* Pregnancy
* Serious internistic diseases
* Drug addiction

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2013-03; Primary Completion 2014-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
pathological comparative results and all cause mobidity | 1 year
  The comparison of these two methods to show that the pathologic diagnostical results are alike and the morbidity is less.

CONTACTS AND LOCATIONS:
Overall Officials: Achim Schneider, Prof. Dr., MPH, Study Chair — Charité University Berlin, Germany
Locations (1):
- Charité, Berlin, Germany

REFERENCES:
- See also: Related Info — http://frauenklinik.charite.de/en/